CLINICAL TRIAL: NCT00680420
Title: DNA Microarray Analysis of Endoscopic Ultrasound-Guided Fine Needle Aspiration Biopsies to Discriminate Benign From Malignant Pancreatic Lesions
Brief Title: DNA Microarray Study of Pancreas Cancer
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Sarah Rodriguez, Physician, Oregon Health and Science University
Other Study IDs: IRB4191
Record Dates: First submitted 2008-05-16; First posted 2008-05-20 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Pancreas Cancer
Keywords: pancreas cancer; pancreas cyst; DNA microarray
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic Cyst | interventions — Biopsy, Fine-Needle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: fine needle aspiration biopsy — One extra biopsy will be taken from the pancreas only in patients who are already undergoing biopsy of a mass or cyst.

SUMMARY:
Pancreas cancer and precancerous cysts can be difficult to diagnose. Sometimes biopsies do not show cancer when cancer is actually present. We hypothesize that genetic differences exist in tissue that is malignant compared to nonmalignant. When patients present with a pancreas mass or cyst, we biopsy it by fine-needle aspiration during upper endoscopy with ultrasound guidance. We would like to use tissue obtained via endoscopic ultrasound guided fine needle aspiration to perform DNA microarray analysis, and compare the differences in gene expression level in the benign tissue compared to cancerous tissue in order to improve our diagnostic capabilities. DNA microarray measures gene expression level rather than germline mutations. The true diagnosis will be based on cytology, surgical pathology, or clinical followup. The performance of the microarray test as a diagnostic test will be compared to the performance of cytology.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 or older who are able to give informed consent who present for an endoscopic ultrasound to evaluate a pancreas mass or cyst or for suspicion of cancer.

Exclusion Criteria:

* Unable to give informed consent, pregnant or nursing, contraindication to endoscopic ultrasound, no mass or cyst found on ultrasound

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with suspected pancreas mass
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2008-06; Primary Completion 2010-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Gene expression profile is 95% accurate in diagnosis of malignancy | after enrollment of 50 patients

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Rodriguez, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States